CLINICAL TRIAL: NCT07166393
Title: Multi-institutional Phase 2/3 Trial of Valproic Acid in Patients With Moderate to Severe Traumatic Brain Injury
Brief Title: Valproic AcId for Traumatic BRAin INjury Trial
Acronym: VIBRANT
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hasan Alam, Chair, Department of Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00223546; HT9425-24-1-0241 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Moderate Traumatic Brain Injury (TBI); Severe Traumatic Brain Injury
Keywords: TBI, traumatic brain injury, VPA, valproic acid
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Valproic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Standard of Care + Normal Saline (0.9% sodium chloride solution)
  Interventions: Other: Standard of care treatment + normal saline
- Experimental (Experimental): Standard of care treatment + one dose of VPA (in 250 ml 0.9% sodium chloride solution) in the following two doses:
  * Lower dose VPA: 50 mg/kg
  * Higher dose VPA: 100 mg/kg
  Interventions: Drug: Valproic Acid (VPA)

INTERVENTIONS:
Drug: Valproic Acid (VPA) — VPA (in 250 ml 0.9% sodium chloride solution)
  Arms: Experimental
Other: Standard of care treatment + normal saline — Standard of care treatment + normal saline (0.9% sodium chloride solution) vehicle (250 ml)
  Arms: Control

SUMMARY:
The long-term goal of the clinical trial is to develop effective, safe, and easily administered life-saving treatments for patients with moderate to severe traumatic brain injury (TBI).

Patients with moderate to severe TBI will randomly receive either:

1. Standard of care treatment and normal saline
2. Standard of care treatment and one dose of valproic acid (VPA) at a lower dose or a higher dose

DETAILED DESCRIPTION:
The specific aim is to determine whether giving VPA at either a 50 mg/kg dose or a 100 mg/kg is safe (as measured by adverse events after treatment) in patients with moderate to severe TBI due to brain bruises.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 65 years.
2. Body Mass Index between 18 kg/m2 and 35 kg/m2.
3. Females must be surgically sterilized, postmenopausal, or have a negative urine pregnancy test.
4. Moderate to severe TBI: Glasgow Coma Scale (GCS) 3-12.
5. Cerebral trauma confirmed on the initial CT scan with radiographic findings consistent with Brain Injury Guidelines category 3 (BIG3) criteria

Exclusion Criteria:

1. Persons with known history of adverse reactions to VPA
2. Persons with known history of hepatitis B or C or clinical history of hepatic dysfunction, pancreatitis, or renal insufficiency.
3. Persons with a known history of thrombocytopenia.
4. Persons with platelet count less than 100,000 per microliter of blood.
5. Persons with 2nd or 3rd degree burns of any size and location.
6. Female subjects who are pregnant or lactating.
7. Persons who are currently incarcerated or are in police custody.
8. Persons with inadequate venous access.
9. Treatment cannot start within 120 minutes from the onset of injury
10. Non-survivable injuries in the estimation of the attending trauma surgeon.
11. Interfacility transfers
12. The time of injury is unknown
13. Patients in hemorrhagic shock with a systolic blood pressure of <90 mmHg on initial evaluation.
14. Persons with a known "do not resuscitate" order prior to randomization
15. Persons with a research "opt out" bracelet
16. Persons who are currently enrolled in another clinical trial.
17. Greater than 90 minutes between the onset of injury and arrival to the hospital

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Extended Glasgow Outcome Scale (GOS-E) | 3 months post-injury
  Scoring values range from 1 to 8 with higher scores representing a better outcome. 1 indicates death, 2 indicates a vegetative state, 3 or 4 indicates severe disability, 5 or 6 indicates moderate disability, and 7 or 8 indicates good recovery.

SECONDARY OUTCOMES:
Hemorrhagic progression of the contusion (HPC) | First 24 hours post-injury as measured by a CT scan
  We will quantify HPC as the change in volume of the largest contiguous brain lesion in mm. This will be measured through a comparison of the initial and the follow-up CT scan.
Disability Rating Score (DRS) | Discharge or day 7 and 3 months post-injury
  This scale includes eight categories: A. Eye opening (0-5), B. Communication ability (0-4), C. Motor response (0-5), D. Feeding - cognitive ability only (0-3), E. Toileting - cognitive ability only (0-3), F. Grooming - cognitive ability only (0-3), G. Level of functioning - physical, mental, emotional or social function (0-5) and H. "Employability" - a full time worker, homemaker, or student (0-3). Higher scores in each category mean a worse outcome.

OTHER OUTCOMES:
Disability Rating Score (DRS) | 6 months post-injury
  This scale includes eight categories: A. Eye opening (0-5), B. Communication ability (0-4), C. Motor response (0-5), D. Feeding - cognitive ability only (0-3), E. Toileting - cognitive ability only (0-3), F. Grooming - cognitive ability only (0-3), G. Level of functioning - physical, mental, emotional or social function (0-5) and H. "Employability" - a full time worker, homemaker, or student (0-3). Higher scores in each category mean a worse outcome.
Extended Glasgow Outcome Scale (GOS-E) | 6 months post injury
  Scoring values range from 1 to 8 with higher scores representing a better outcome. 1 indicates death, 2 indicates a vegetative state, 3 or 4 indicates severe disability, 5 or 6 indicates moderate disability, and 7 or 8 indicates good recovery.
Glasgow Coma Scale (GCS) | 24 hours post-injury
  Evaluates three behavior responses: eye opening, best verbal and best motor. The following scoring is associated with responses: Eye opening response - Spontaneously 4, To speech 3, To pain 2 and No response 1; Best verbal - Oriented to time/place/person 5, Confused 4, Inappropriate words 3, Incomprehensible sounds 2 and No response 1; and Best motor response - Obeys commands 6, Moves to localized pain 5, Flexion withdrawal from pain 4, Abnormal flexion 3, Abnormal extension 2 and No response 1. The scoring is totaled with higher values associated with better response. Total Score: Best response=15, Comatose client=8 or less, and Totally unresponsive=3.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Alam, MD, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared.

REFERENCES:
- [Derived] Visa MA, Liggett MR, Lashley S, Bhatti U, Dawood ZA, Anand A, Gill NP, Scholtens DM, Wang B, Alam HB. Valproic acid for treatment of traumatic brain injury: Study protocol for the VIBRANT prospective randomized trial. Transfusion. 2025 Dec 20. doi: 10.1111/trf.70029. Online ahead of print. PMID 41420823